CLINICAL TRIAL: NCT04165161
Title: Performance Diagnosis of a Patent Foramen Ovale During Lung Transplantation Using Transesophageal Echocardiography: Comparison of the Injection of Contrast in the Upper and Lower Caval Territories (FOP-TP)
Brief Title: Performance Diagnosis of a Patent Foramen Ovale During Lung Transplantation Using Transesophageal Echocardiography
Acronym: FOP-TP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018_0098
Record Dates: First submitted 2019-10-29; First posted 2019-11-15 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Lung Transplant; Complications

STUDY DESIGN:
Intervention Model Description: For each patient the 4 tests will be performed in a randomized order to limit bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- superior without positive tele-expiratory pressure (Other): Diagnostic Test: Contrast injection in the superior vena cava territory + controlled ventilation without positive tele-expiratory pressure
  Interventions: Diagnostic Test: search for a patent foramen ovale
- superior with 10 cmH2O positive tele-expiratory pressure (Other): Diagnostic Test: Contrast injection in the superior vena cava territory + controlled ventilation with 10 cmH2O positive tele-expiratory pressure
  Interventions: Diagnostic Test: search for a patent foramen ovale
- inferior without positive tele-expiratory pressure (Other): Diagnostic Test: Contrast injection in the inferior vena cava territory + controlled ventilation without positive tele-expiratory pressure
  Interventions: Diagnostic Test: search for a patent foramen ovale
- inferior with 10 cmH2O positive tele-expiratory pressur (Other): Diagnostic Test: Contrast injection in the inferior vena cava territory + controlled ventilation with 10 cmH2O positive tele-expiratory pressure
  Interventions: Diagnostic Test: search for a patent foramen ovale

INTERVENTIONS:
Diagnostic Test: search for a patent foramen ovale — Injection of a contrast solution A - In the upper cellar territory with controlled ventilation without positive tele-expiratory pressure; B - In the upper cellar territory in controlled ventilation with a positive end-to-expiratory pressure of 10cm H2O; C - In the lower cellar territory with controlled ventilation without positive tele-expiratory pressure; D - In the lower cellar territory in controlled ventilation with a positive end-to-expiratory pressure of 10cm H2O;

SUMMARY:
The investigators hypothesis is that an injection into the inferior vena cava associated with a provocation maneuver should allow to increase the incidence of FOP found by transesophageal echocardiography in a population of patients undergoing lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old minimum
* Benefiting from a lung transplant
* Having an upper vena cava catheter and a lower vena cava catheter set up as part of the usual care
* Having signed a consent form
* Affiliated to a insurance scheme or beneficiary (excluding AME)

Exclusion Criteria:

* Pregnant or lactating women
* Having a contraindication to the insertion of the esophageal ultrasound probe
* deprived of liberty or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of transatrial passage of contrast media | 1 day after lung transplantation
  Incidence of transatrial passage of contrast media

SECONDARY OUTCOMES:
Size of PFO, existence of an atrial septal aneurysm | 1 day after lung transplantation
Number of postoperative days with mechanical ventilation | 30 days after lung transplantation
Incidence of pulmonary graft dysfunction, incidence of stroke, incidence of myocardial ischemia | 30 days after lung transplantation
Mortality during the stay in the intensive care unit | 30 days after lung transplantation
Mortality during the stay in the hospital | 30 days after lung transplantation
Mortality at the postoperative 30-day | 30 days after lung transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Davignon, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France